CLINICAL TRIAL: NCT03288597
Title: A Prospective Exploration in the Clinical Value of 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT in Neuroendocrine Neoplasms
Brief Title: Explore the Clinical Value of 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT in Neuroendocrine Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Other Study IDs: 68Ga&FDG PET/CT
Record Dates: First submitted 2017-09-16; First posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Neuroendocrine Tumors
Keywords: positive rate; SUVmax; relationship
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: advanced and metastatic neuroendocrine tumors: Advanced and metastatic neuroendocrine tumors receive syestematic treatment
  Interventions: Radiation: 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT in NET
- A: advanced and metastatic neuroendocrine carcinomas: Advanced and metastatic neuroendocrine carcinomas receive syestematic treatment
  Interventions: Radiation: 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT in NEC

INTERVENTIONS:
Radiation: 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT in NET — At the beginning of the treatment with SSA, after 6 months, 12 months, or chemotherapy, after 3 months or progression receive 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT
  Groups: A: advanced and metastatic neuroendocrine tumors
Radiation: 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT in NEC — At the beginning of the treatment with chemotherapy 4-6 cycles or progression receive 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT
  Groups: A: advanced and metastatic neuroendocrine carcinomas

SUMMARY:
68Ga-DOTANOC and 18F-FDG PET/CT have important values in the staging and clinical treatment of neuroendocrine tumors. Retrospective studies suggest that the positivite rates and SUVmax of dual imaging associated with pathological findings and prognosis. The study was designed to confirm thet clinical values of dual imagings for neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. sign written informed consent form
2. age ≥ 18 years
3. pathologically confirmed neuroendocrine, Ki67>=10%;
4. ECOG 0-1;
5. No prior antitumor treatment with chemotherapy targeting regimens for neuroendocrine carcimomas, no more than 2 systematic treatment for neuroendocrine tumors;
6. Unresectable disease;
7. At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions);
8. Predicted survival >=3 months;
9. Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women;
10. Sexually active males or females willing to practice contraception during the study until 30 days after end of study.

Exclusion Criteria:

1. In the process of antitumor therapy with effective response;
2. Refuse to accept PET/CT;
3. Pregnant or nursing, or sexually active males or females refuse to practice contraception during the study until 30 days after end of study;
4. Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Neuroendocrine neoplasmes
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between the positive rate and SUVs of 68Ga-DOTANOC PET/CT and 18F-FDG PET/CT and treatment response | 3 years

SECONDARY OUTCOMES:
The correlation between positive rate and SUV of PET/CT and prognosis | 3 year
Compare SUVmax, tumor/liver ratio as a prognostic marker | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No